CLINICAL TRIAL: NCT05700214
Title: Continuous Infusion of Lidocaine Versus Blockade of the Erector Spinae Plane Block - Comparison of Analgesic Efficacy in Patients After Bariatric Surgery
Brief Title: Lidocaine Versus ESP - After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, Principal Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1072.6120.249.2022
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Anesthetics; Local Anesthetics
Keywords: Acute Pain; Pain; Ropivacaine; Anesthetics, Local; Physiological Effects of Drugs
MeSH Terms: conditions — Acute Pain; Pain | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESP block (Experimental): Ultrasound-guided continuous ESP block with opioid PCA A high-frequency linear ultrasound transducer will be placed in a longitudinal parasagittal orientation 3 cm lateral to the T7/T8 spinous process. A Contiplex Echo ultra 360 18G needle with 20G × 55 cm Contiplex Echo catheter will be inserted using an in-plane superior-to-inferior approach to place the tip into the fascial plane on the deep (anterior) aspect of erector spinae muscle. The location of the needle tip will be confirmed by visible fluid spread lifting erector spinae muscle off the bony shadow of the transverse process. A total of 30 mL of 0.35% ropivacaine
  Interventions: Drug: Ropivacaine injection
- lidocaine (Active Comparator): Before induction bolus of 1% lidocaine 1,5mg/kg IBW i.v., continuous infusion of 1% lidocaine intraoperatively rate 1 mg/kg IBW i.v.
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Ropivacaine injection — 30ml of 0.35% ropivacaine
  Other Names: ESP block
  Arms: ESP block
Drug: Lidocaine IV — Before induction bolus of 1% lidocaine 1,5mg/kg IBW i.v., continuous infusion of 1% lidocaine intraoperatively rate 1 mg/kg IBW i.v.
  Other Names: Lidocaine infusion
  Arms: lidocaine

SUMMARY:
The Erector Spinal Block (ESP) is based on the deposition of the local anesthetic in the inter-fascial space between the dorsal extensor muscle and the intercostal muscles at the height of the transverse processes. The scope of the blockade covers the dorsal and ventral branches of the thoracic spinal nerves, but also in most cases the investigetors are able to obtain a wide distribution of the drug into the paravertebral space by "permeating" the local anesthetic through the fascial compartments. The clinical effect of the blockade is due to blocking the nerve structures of the paravertebral space (spinal nerve branches and the sympathetic trunk). The scope of the blockade, after its execution at the level of Th5, most often includes the segments from Th1 to L1.

Lidocaine used in intravenous infusion is one of the recommended components of multidirectional analgesia. Its adjuvant properties make it possible to reduce the amount of opioid drugs used, and thus - to reduce the frequency of their side effects.

The aim of the study is to test the effectiveness and safety of the use of lidocaine infusion or Erector Spinal Block in multimodal analgesic management.

DETAILED DESCRIPTION:
In bariatric surgery, overall pain is a conglomerate of three different and clinically separate components: incisional pain (somatic pain), visceral pain (deep intra abdominal pain), and shoulder pain due to peritoneal stretching and diaphragmatic irritation associated with carbon dioxide insufflation. Moreover, it has been hypothesized that intense acute pain after labdomen surgery may predict development of chronic pain. Without effective treatment, this ongoing pain may delay recovery, mandate inpatient admission, and thereby increase the cost of such care.

ELIGIBILITY:
Inclusion Criteria:

Patients requiring bariatric surgery Obesity (BMI>35)

Exclusion Criteria:

Patient refusal Contraindications to paravertebral blocks: Infection at the site of needle insertion, empyema, allergy to local anesthetic drugs, and tumor occupying the thoracic paravertebral space, coagulopathy, bleeding disorder or therapeutic anticoagulation Known allergy to local anesthetics Inability to provide informed consent Any patient on opioids for greater than or equal to 3 months duration prior to surgery Patients with chronic pain syndromes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Total long acting opioid consumption in oxycodone equivalents | 1 day
  the total dosage of given drug
Pain scores will be recorded at intervals. | 1 days
  The Numerical Rating Scale (NRS) is an 11-point scale where 0 is no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Skladzien, MD PHD, Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No